CLINICAL TRIAL: NCT04979065
Title: Effect of Probiotic and Vitamin D Supplementation in Modulating Gut Dysbiosis, Nutrition, Inflammation and Immune Status and Reduce Risk of COVID-19 in Obese People: Gut-Lung Axis Randomized Trial
Brief Title: Nutrition, Immunity, and Covid-19 in Obese People
Acronym: NICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, Head of Human Nutrition Research Centre / Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICO
Record Dates: First submitted 2021-07-24; First posted 2021-07-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Vitamin D Deficiency; Covid19; Overweight and Obesity; Immune Deficiency
Keywords: Probiotics; Vitamin D; Immune status; Covid-19; Nutrition
MeSH Terms: conditions — Vitamin D Deficiency; COVID-19; Overweight; Obesity; Immunologic Deficiency Syndromes | interventions — Probiotics; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Independent party masked the intervention and control product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Probiotics and Vitamin D
  Interventions: Dietary Supplement: Probiotics, Vitamin D
- Control Group (Placebo Comparator): Placebo and placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics, Vitamin D — Combination of two supplement that given separately
  Arms: Experimental Group
Other: Placebo — Placebo with inactive ingredient
  Arms: Control Group

SUMMARY:
The increased risk of transmission of COVID-19 infection causes the incidence of death in health workers to escalate. It requires further research on risk factors and intervention in health worker professionals, especially on immunity factors and nutritional status. Quality of diet and nutrition is very important to support the immune system when infected. Several probiotic strains have been shown to decrease the duration and incidence of diarrhea and respiratory infections, suggesting the Gut-Lung Axis pathway. Some probiotics also improve the balance of diversity in the composition of the gut microbiota and affect body weight in obese people. Probiotics have also been shown to improve vitamin D absorption. A combination of vitamin D and probiotics may be an alternative to reduce gut dysbiosis that will directly or indirectly reduce the risk and severity of viral infections including SARS-CoV-2.

DETAILED DESCRIPTION:
Obesity is increasing in Indonesia and is the cause of various diseases, especially in the presence of Vitamin D deficiency, a state of dysbiosis, causing an increase in the possibility of infection. Professional health workers have a high risk of COVID-19 due to high daily exposure. Based on a review conducted by Daniel et al, it was found that 7.3% of health workers at Reutters University tested positive for COVID-19. Based on data from the Indonesian Doctors Association (IDI) on July 12, 2020, it was known that 61 doctors had died. In addition, based on data from the Indonesian National Nurses Association (PPNI), 39 nurses have died during the COVID-19 pandemic. Therefore efforts to prevent the occurrence of COVID-19 infection by providing a combination of vitamin D and probiotics to modulate dysbiosis that will further reduce the risk of viral infection, especially COVID-19, needs to be investigated for its potential benefits.

Primary and secondary objectives

1. Primary Objective:

   To investigate the effect of a combination of probiotics and vitamin D supplementation in modulating intestinal dysbiosis, and vitamin D status, in people with overweight and obesity, especially among frontline health workers.
   * To assess the mean changes in zonulin levels (as a parameter of gut integrity to indicate the intestinal microbiota dysbiosis)
   * To assess the mean changes in serum vitamin D levels
2. Secondary Objectives:

   * To assess the relationship between nutritional status, inflammation and immunity with the risk of COVID-19 infection in health workers.
   * To understand the difference in the mean episodes of Covid-19 infection between treatment and placebo groups after giving probiotics and vitamin D in people with overweight and obesity, especially among frontline health workers.

Study Design:

This study has 2 phases Phase 1: a Cross-sectional study with 160 people Phase 2: a double-blind, randomized, placebo-controlled trial with two arms of intervention involving a total of 80 people.

ELIGIBILITY:
Inclusion Criteria:

* General doctors, specialist doctors, nurses and midwives who are in charge of handling COVID-19 patients or working in COVID-19 referral hospitals for at least the last 3 months
* 20-65 years old
* Willing to sign informed consent
* Willing to follow the research to completion
* BMI > 23 kg/m2

Exclusion Criteria:

* Pregnant woman
* Have a confirmed history of COVID-19 based on previous PCR examinations
* Suffering from acute illness known from history and physical examination or chronic disease (eg diabetes, SLE, cardiovascular disease) known from history
* Currently not on a diet program for weight loss or consuming probiotics regularly in the last 3 months as known from the anamnesis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Zonulin level | Baseline and endline (3 month)
  To investigate the changes of Zonulin level during intervention
Vitamin D level | Baseline and endline (3 month)
  To investigate the changes of Vitamin D level during intervention

SECONDARY OUTCOMES:
Nutritional status | Baseline and endline (3 month)
  Measurement of nutritional status using Body Mass Index (BMI) and waist circumference
Gut microbiota (optional) | Baseline and endline (3 month)
  Measurement of gut microbiota in fecal using Next Generation Sequencing
Inflammation marker | Screening
  Measurement of inflammation markers IL-6, IL-10 TNF-α using ELISA
Cathelicidin level | Screening
  Measurement of cathelicidin using ELISA
SARS COV-2 | Screening
  Measurement of quantitative antibody
CD4/CD8 ratio | Screening
  Measurement of CD4/CD8 ratio using flowcytometry
Covid-19 infection | Baseline and endline (3 month)
  Measurement of the reduction in risk of COVID-19 infection is seen from the difference in the average episodes between groups that were examined by PCR and/or Rapid antibody tests.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, MD, PhD, Principal Investigator — HNRC-IMERI, Faculty of Medicine Universitas Indonesia
Locations (4):
- Indonesia (4):
  - Wisma Emergency COVID-19 Hospital (RSDC), Jakarta, DKI Jakarta
  - Department of Nutrition (FKUI-RSCM); and Human Nutrition Research Center, Indonesian Medical Education Research Institute (HNRC-IMERI) Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta
  - Dr.Cipto Mangunkusumo General Hospital (RSCM), Jakarta Pusat, DKI Jakarta
  - University of Indonesia Hospital (RSUI), Depok, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong NS, Zheng BJ, Li YM, Poon, Xie ZH, Chan KH, Li PH, Tan SY, Chang Q, Xie JP, Liu XQ, Xu J, Li DX, Yuen KY, Peiris, Guan Y. Epidemiology and cause of severe acute respiratory syndrome (SARS) in Guangdong, People's Republic of China, in February, 2003. Lancet. 2003 Oct 25;362(9393):1353-8. doi: 10.1016/s0140-6736(03)14630-2. PMID 14585636
- [Background] Shereen MA, Khan S, Kazmi A, Bashir N, Siddique R. COVID-19 infection: Origin, transmission, and characteristics of human coronaviruses. J Adv Res. 2020 Mar 16;24:91-98. doi: 10.1016/j.jare.2020.03.005. eCollection 2020 Jul. PMID 32257431
- [Background] Sattar N, McInnes IB, McMurray JJV. Obesity Is a Risk Factor for Severe COVID-19 Infection: Multiple Potential Mechanisms. Circulation. 2020 Jul 7;142(1):4-6. doi: 10.1161/CIRCULATIONAHA.120.047659. Epub 2020 Apr 22. No abstract available. PMID 32320270
- [Background] Kass DA, Duggal P, Cingolani O. Obesity could shift severe COVID-19 disease to younger ages. Lancet. 2020 May 16;395(10236):1544-1545. doi: 10.1016/S0140-6736(20)31024-2. Epub 2020 May 4. No abstract available. PMID 32380044
- [Background] Nagpal R, Newman TM, Wang S, Jain S, Lovato JF, Yadav H. Obesity-Linked Gut Microbiome Dysbiosis Associated with Derangements in Gut Permeability and Intestinal Cellular Homeostasis Independent of Diet. J Diabetes Res. 2018 Sep 3;2018:3462092. doi: 10.1155/2018/3462092. eCollection 2018. PMID 30250849
- [Background] Calder PC, Carr AC, Gombart AF, Eggersdorfer M. Optimal Nutritional Status for a Well-Functioning Immune System Is an Important Factor to Protect against Viral Infections. Nutrients. 2020 Apr 23;12(4):1181. doi: 10.3390/nu12041181. PMID 32340216
- [Background] Childs CE, Calder PC, Miles EA. Diet and Immune Function. Nutrients. 2019 Aug 16;11(8):1933. doi: 10.3390/nu11081933. PMID 31426423
- [Background] Wong SH, Lui RN, Sung JJ. Covid-19 and the digestive system. J Gastroenterol Hepatol. 2020 May;35(5):744-748. doi: 10.1111/jgh.15047. Epub 2020 Apr 19. PMID 32215956
- [Background] King S, Glanville J, Sanders ME, Fitzgerald A, Varley D. Effectiveness of probiotics on the duration of illness in healthy children and adults who develop common acute respiratory infectious conditions: a systematic review and meta-analysis. Br J Nutr. 2014 Jul 14;112(1):41-54. doi: 10.1017/S0007114514000075. Epub 2014 Apr 29. PMID 24780623